CLINICAL TRIAL: NCT03175107
Title: mHealth Platform for Parkinson's Disease Management: Exergaming in Upper Extremities for Persons With Parkinson's Disease
Brief Title: Exergaming in Upper Extremities for Persons With Parkinson's Disease
Acronym: PD_managerSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Collaborators: Jozef Stefan Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: URIS201702
Record Dates: First submitted 2017-05-22; First posted 2017-06-05 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Parkinson Disease
Keywords: exergaming; physiotherapy; upper extremities; telerehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD_patients (Experimental): Patients with Parkinson disease or Parkinsonism (characteristic symptoms such as rigidity, extrapyramidal symptoms), with functional disorders in upper extremities and minor problems at daily activities, with the level 2-3 in the Hoehn and Yahr Scale. They will perform exergaming at home for up to 4 weeks.
  Interventions: Device: Exergaming

INTERVENTIONS:
Device: Exergaming

SUMMARY:
The purpose of the PD_manager project is to explore and develop innovative ecosystem management for people with Parkinson's disease. The research part contains expert analysis of diagnostic tests and decomposition of activity, accompanied by modern IT. The results of the analysis will be compared with the results of clinical trials that fall under the routine clinical pathways in monitoring a patient with Parkinson's disease. The primary motor symptoms, such as tremor, bradykinesia and impaired balance, and other symptoms, such as sleep disturbances, speech and cognitive perception, will be assessed by unobtrusive sensors (shoe insoles, bracelets) and sensors embedded in a mobile phone. The collected data will be analyzed using data mining methods and a platform for clinical decision support will be developed. This way, dependency of the patients on other persons will be reduced and the patients' quality of life improved. The patients will be motivated to follow the prescribed diet and take regular medication; the patients' activities will be monitored by occupational therapists and physiotherapists. A technical system will be designed as a computing platform in the open architecture cloud (FI-WARE), which will allow the use of commercially available sensors.

DETAILED DESCRIPTION:
The application of tasks in virtual reality and computer games for motoric exercise in patients with neurologic impairment is already quite widespread. It allows controlled workout and flexible gradation of difficulty of the task, which is essential for rehabilitation. Even in patients with Parkinson's disease, it allows for the gradual physiotherapy to improve range of mobility and improve fine motor skills of upper extremities. Within the project, existing games (Microsoft Xbox, Kinect) will be used and a special application for the Microsoft Kinect and Leap Motion systems will be developed, both for the movement of upper extremities as well as fine motor skills (plugs, 9 hole, labyrinth). Both systems will allow data storage, overview of the results, and the algorithm will also adapt the difficulty level of the tasks. This will allow creation of scenarios, as well as monitoring the gradual progress in rehabilitation. The study will begin with treatment in a hospital (URI-Soca), testing three platforms (Kinect, Leap Motion, plate). The most appropriate and most scalable solution will be further developed to the stage where it can be installed in the patient's home. The control of the system and data access will be performed remotely via the Internet and/or mobile phone. When the system is tested and evaluated at the patient's home, a user-friendly application will be developed for the patient to set the desired functions, for the therapist to set difficulty levels and provide instructions to the patient, and for the physician to examine the data and clinically evaluate the patient's condition.

The participants will test the application for up to 4 weeks and then report on the user experience. A standardized questionnaire (NRS 2002) will be used for this purpose. URI-Soca will recruit at least 7 patients, inpatients or outpatients for motor rehabilitation of upper extremities. The tasks will be carried out at the occupational therapy and physiotherapy units of URI-Soca for up to 4 weeks, 3 times a week. At the same time, expert analysis (neurologist, physiotherapist, occupational therapist, engineer) of the measured data (kinematics, the results achieved) will be performed and clinical tests (Unified Parkinson's Disease Rating Scale - UPDRS, Jebsen Tailor Functional Test and PD Questionnaire 39) will be carried out before and after the exercise program. At the same time, the system will be adapted for home use (by at least 1 patient), and then a study will be conducted with other patients. These participants will receive the system for home use for up to 60 days. The data will be accessed remotely over the Internet, so the objective evaluation can be carried out promptly. The clinical test will be conducted before exercise and after exercise, i.e., at the beginning and at the end of the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease or Parkinsonism (characteristic symptoms such as rigidity, extrapyramidal symptoms), with functional disorders in upper extremities and minor problems at daily activities;
* Level 2-3 in the Hoehn and Yahr Scale.

Exclusion Criteria:

* Any communicable disease;
* Severe vision impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Box & Blocks Test from baseline | Assessment at baseline and at five weeks
  Standard clinical test to assesses unilateral gross manual dexterity

SECONDARY OUTCOMES:
Change in Nine Hole Peg Test from baseline | Assessment at baseline and at five weeks
  Standard clinical test for measuring finger dexterity and other aspects of upper extremity function
Change in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) from baseline | Assessment at baseline and at five weeks
  MDS-UPDRS is a comprehensive assessment designed to monitor the burden and extent of Parkinson's disease
Change in Jebsen Hand Function Test (JHFT) from baseline | Assessment at baseline and at five weeks
  JHFT assesses a broad range of uni-manual hand functions required for activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Imre Cikajlo, PhD, Principal Investigator — University Rehabilitation Institute, Rehabilitation of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cikajlo I, Hukic A, Zajc D. Exergaming as Part of the Telerehabilitation Can Be Adequate to the Outpatient Training: Preliminary Findings of a Non-randomized Pilot Study in Parkinson's Disease. Front Neurol. 2021 Mar 16;12:625225. doi: 10.3389/fneur.2021.625225. eCollection 2021. PMID 33815252